CLINICAL TRIAL: NCT03701568
Title: A RETROspective Study of the Combination of Pyrimidine Nucleos(t)Ides in Patients With Thymidine Kinase 2 Deficiency (TK2)
Brief Title: A RETROspective Study of Patients With TK2d
Acronym: RETRO
Status: Completed | Type: Observational
Sponsor: Zogenix MDS, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: MT-1621-101
Record Dates: First submitted 2018-09-27; First posted 2018-10-10 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Thymidine Kinase 2 (TK2)
Keywords: myopathy, muscle weakness, hypotonia, dysphagia, ptosis
MeSH Terms: conditions — Muscular Diseases; Muscle Weakness; Muscle Hypotonia; Deglutition Disorders; Blepharoptosis | interventions — Deoxycytidine; Thymidine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — When available, test reports maybe obtained (eg, reports from genetic testing, muscle biopsy) as well as available research biological samples (eg, blood or tissue samples that may be tested for biomarkers of disease and/or effects of medications to treat the mitochondrial disease).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: dC/dT — Collection of retrospective data from TK2 patients previously treated with dC/dT
  Other Names: deoxycytidine/deoxythymidine

SUMMARY:
This is a medical chart review study to collect information for patients who have been taking pyrimidine nucleosides for treatment of TK2 deficiency. Information from the time of onset of symptoms will be collected to describe the pre treatment course of TK2 deficiency.

DETAILED DESCRIPTION:
Data to be collected from the time of onset of symptoms related to TK2 deficiency includes medical conditions and/or adverse events (AEs); these should include relationship to TK2 disease and/or pyrimidine nucleosides, as appropriate, as well as date of onset and severity, when available. When available, test reports may be obtained as well as available research biological samples (eg, blood or tissue samples that may be tested for biomarkers of disease and/or effects of medications to treat the mitochondrial disease).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the patient or parent(s)/legally authorized representative (LAR) and/or assent by the patient (when applicable), unless the associated institutional review board (IRB) or ethics committee (EC) provides an appropriate consent waiver
2. Confirmed genetic mutation in the TK2 gene
3. Availability of medical records for each patient from the time of onset of symptoms
4. Patient has taken pyrimidine nucleos(t)ides (dCMP/dTMP and/or dC/dT) as substrate enhancement therapy for TK2 deficiency
5. Most recent patient visit at which efficacy and/or safety parameters were collected occurred between 01 June 2018 and 15 December 2018

Exclusion Criteria:

1. Presence of other genetic disease or polygenic disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with TK2 deficiency who have received treatment with pyrimidine nucleosides
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnosis | 3 months
  genetic testing (previously conducted)

SECONDARY OUTCOMES:
Clinical course | 3 months
  BMI (height in inches and weight in kg will be combined to report BMI in kg/m^2)
Clinical course | 3 months
  achievement, loss, or regaining of developmental motor milestones
Motor function and ambulatory assessments | 3 months
  Change in 6-minute walk test [6MWT] distance (in meters)
Motor function and ambulatory assessments | 3 months
  Motor Function Measure [MFM] 20 or MFM 32
Motor function and ambulatory assessments | 3 months
  Egen Klassifikation
Motor function and ambulatory assessments | 3 months
  North Star Ambulatory Assessment
Motor function and ambulatory assessments | 3 months
  Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders [CHOP INTEND]
Motor function and ambulatory assessments | 3 months
  Hammersmith Functional Motor Scale-Expanded [HFMSE]

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (8):
- Columbia University Medical Center, New York, New York, United States
- Israel (3):
  - Rambam Hospital, Haifa
  - Wolfson Medical Center, Holon
  - Western Galilee Hospital, Nahariya
- Spain (4):
  - Hospital Vall d'Hebron, Barcelona
  - Sant Joan de Déu Hospital, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dominguez-Gonzalez C, Chiang C, Colson AO, Rebollo Mesa I, Baixauli E, Quan J, VanMeter S, Hirano M. Pyrimidine Nucleos(t)ide Therapy in Patients With Thymidine Kinase 2 Deficiency: A Multicenter Retrospective Chart Review Study. Neurology. 2025 Sep 23;105(6):e213908. doi: 10.1212/WNL.0000000000213908. Epub 2025 Sep 5. PMID 40911819